CLINICAL TRIAL: NCT05143762
Title: Effect of Preemptive Dexamethasone and Paracetamol on Postoperative Period Following Adeno-tosillectomy in Pediatric Age Group-: A Randomized Clinical Trial
Brief Title: Preemptive Dexamethasone , Paracetamol on Postoperative Period Following Adeno-tonsillectomy in Pediatric .
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-10-2021
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Analgesia
Keywords: analgesia; dexamethasone; paracetamol
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group (A) (Active Comparator): will receive intravenous paracetamol 30mg/kg (max 90 mg/kg/day).
  Interventions: Drug: paracetamol
- group (B) (Active Comparator): will receive dexamethasone 0.5mg/kg IV.
  Interventions: Drug: Dexamethasone
- group(C) (Placebo Comparator): will received placebo 10 ml normal saline IV.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: paracetamol — patients will receive intravenous paracetamol 30mg/kg (max 90 mg/kg/day)
  Arms: group (A)
Drug: Dexamethasone — patients will receive dexamethasone 0.5mg/kg IV.
  Arms: group (B)
Drug: normal Saline — patients will receive placebo 10 ml normal saline IV.
  Arms: group(C)

SUMMARY:
Tonsillectomy is one of the most common surgical operations performed on children, and it is frequently linked with an increased risk of complications such as acute discomfort when swallowing and postoperative nausea and vomiting (PONV).The most prevalent causes for postponing discharge home are poorly managed pain and PONV.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common surgical operations performed on children, and it is frequently linked with an increased risk of complications such as acute discomfort when swallowing and postoperative nausea and vomiting (PONV). The most prevalent causes for postponing discharge home are poorly managed pain and PONV. As a result, these occurrences should be avoided and managed utilizing a multimodal strategy Because of its low cost and adequate safety profile in the treatment of post-tonsillectomy pain, acetaminophen is presently regarded the fundamental analgesic in this situation. Furthermore, acetaminophen has been recommended for use in children, and its pharmacological safety in this age group has been shown. Dexamethasone is another medication that is used to reduce postoperative pain and PONV in various procedures.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 3 and 16 years.
* All patients are ASA physical status I or II scheduled to undergo a tonsillectomy with or without adenoidectomy using sharp dissection technique.

Exclusion Criteria:

* psychiatric illness.
* cardiac disease.
* renal or hepatic impairment.
* allergy dexamethasone , paracetamol and opioids.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption at PACU | two hours postoperatively
  total amount of opioid that will be taken by the patients postoperatively.

SECONDARY OUTCOMES:
objective pain score | at 0 minute , 30 minutes ,1 hour and 2 hours at PACU
  pain score will be assessed by 4 points pain scale 0=no pain 1 = mild pain 2= moderate pain 3=severe pain

CONTACTS AND LOCATIONS:
Overall Officials: fatma ahmed abdelfatah, MD, Principal Investigator — Benha University
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt

IPD SHARING:
Plan to Share IPD: Undecided